CLINICAL TRIAL: NCT05877157
Title: Pain and Opioids After Surgery (PANDOS) Study
Brief Title: Pain AND Opioids After Surgery
Acronym: PANDOS
Status: Recruiting | Type: Observational
Sponsor: University of Aberdeen (Other)
Collaborators: European Society of Anaesthesiology and Intensive Care (Other)
Responsible Party: Sponsor
Other Study IDs: 2-082-21
Record Dates: First submitted 2023-04-06; First posted 2023-05-26 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Opioid Use; Pain, Chronic; Pain, Postoperative; Quality of Life
MeSH Terms: conditions — Chronic Pain; Pain, Postoperative

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to document the perioperative opioid use and its safety in the UK and countries in Europe and to describe its association with surgical complications, persistent pain and quality of life. In an international, prospective, observational cohort study, data about the perioperative pain management will be collected in all eligible hospitalised adult patients who undergo surgery in a designated "study week" in as many hospitals as possible in Europe. Baseline data will be collected, and participants followed up at one week, and at three and twelve months post-operatively. The primary outcome will be opioid use at three months after surgery. Secondary outcomes will include opioid use during the preoperative month (preoperative use), during surgery and up to one week after surgery (or discharge, whichever is earlier), and up to the end of the postoperative year. Additional secondary outcomes are the incidence of preoperative pain, persistent pain with/without the presence of neuropathic components, quality of life and surgical complications. The potential association between opioid use and pain outcomes will be investigated. This study could help to develop strategies to improve quality of care, through pain management, for patients undergoing surgery.

DETAILED DESCRIPTION:
PANDOS is an international, prospective, observational cohort study. In a one week period (the designated "study week"), data will be collected in all eligible hospitalised adult patients who undergo surgery in as many hospitals as possible in the UK and Europe. Participants will be followed up for 12 months

ELIGIBILITY:
Inclusion Criteria:

* hospitalised adult patients (18 years and older) undergoing any inpatient surgery (elective or emergency) during the designated study week where an anaesthetist is involved (general anaesthetic, sedation, local anaesthetic).

Able to understand and has capacity to give written informed consent

Exclusion Criteria:

* American Society of Anaesthesiologists (ASA) grade V or VI
* Refusal to participate.
* Lack of comprehension of validated questionnaires or inability to complete the follow-up for any reason.
* Lack of capacity to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All eligible patients undergoing surgery at the hospital during the designated study week
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Patient reported Opioid use post surgery | 3 months
  Patient reported use of opioids post surgery

SECONDARY OUTCOMES:
Opioid use | From recruitment to 1 year post surgery
  Patient reported use of opioids pre-op and opioids used during surgery and prescribed post surgery
Patient reported incidence of pain pre-op and post surgery using BPI-SF | From recruitment to 1 year post surgery
  Patient reported incidence of pain pre-op and post surgery using BPI-SF
Patient reported incidence of pain pre-op and post surgery using DN2 | From recruitment to 1 year post surgery
  Patient reported incidence of pain pre-op and post surgery using DN2
Surgical complications | During surgery
  Recording of surgical complications during surgery
Participant reported quality of life EQ5D-5L | From recruitment to 1 year post surgery
  EQ5D-5L
Participant reported quality of life BPI-SF | From recruitment to 1 year post surgery
  BPI-SF

CONTACTS AND LOCATIONS:
Overall Officials: Patrice Forget, Principal Investigator — University of Aberdeen
Locations (4):
- Department of Anaesthesiology Sestre Milosrdnice, University Hospital Center, Zagreb, Vinogradska 29, Croatia
- United Kingdom (3):
  - NHS Grampian, Aberdeen
  - University College London Hospitals NHS Foundation Trust, London
  - Kings Mill Hospital, Sherwood Forest Hospitals NHS Foundation Trust, Nottingham

IPD SHARING:
Plan to Share IPD: No